CLINICAL TRIAL: NCT03438175
Title: Randomized, Multicenter, Before-after Study for a Large-scale Evaluation of the Effectiveness of a Multitasking Intervention to Improve the Communication Towards Families of Critically Ill Patients
Brief Title: Intensiva 2.0: Improve the Communication Towards Families of Critically Ill Patients
Acronym: Intensiva2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Collaborators: Catholic University of the Sacred Heart (Other); Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other); Società Italiana di Anestesia, Rianimazione, Emergenza e Dolore (SIARED) (Unknown); Ass. Anestesisti Rianimatori Ospedalieri Italiani - Em. Area Crit. (AAROI-EMAC) (Unknown); Associazione Nazionale Infermieri di Area Critica (ANIARTI) (Unknown)
Responsible Party: Principal Investigator, Giovanni Mistraletti, Confirmed University Researcher / Assistant Professor San Paolo University Hospital, Milan, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35410/2017
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Critical Illness; Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic
Keywords: Post-traumatic Stress Disorder; Web-site; Communication; Intensive Care Unit; Comprehension
MeSH Terms: conditions — Critical Illness; Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Families of Critically Ill will be informed about patients'clinical status only by oral communication during daily family meeting
- Intervention (Experimental): Families of critically ill patients will receive during the first ICU day of their loved one a brochure presenting the ICU and inviting them to visit a website specifically created for this project: www.intensiva.it Moreover, in the waiting room of the ICU will be placed 8 posters to improve comprehension and to legitimize emotions.
  Interventions: Behavioral: Enhanced communication by brochure, website and posters

INTERVENTIONS:
Behavioral: Enhanced communication by brochure, website and posters — Several instruments to improve communication toward ICU patients' families were prepared for this study: a brochure of 12 pages, a website with 80 webpages, 8 posters for the waiting room, 1 sign for the ICU door. All these instruments are made to have more correct comprehension and to legitimize emotions of ICU patients' families.
  Arms: Intervention

SUMMARY:
The admission of a loved one in an ICU is a hard experience for family members. They frequently feel fear and grief, develop anxiety and depression symptoms, or even show some behaviors as this event was a real traumatic one, like hyper-arousal, avoidance and intrusion in the daily life.To improve the communication between them and the ICU staff members, and to meet their needs in terms of medical comprehension and emotional legitimization, a specific website was built, and a brochure was printed to make them welcomed in the ICU; moreover, a series of poster was prepared for the family waiting room outside the ICU. These instruments appeared able to improve the correctness of prognosis comprehension and to decrease the post-traumatic stress symptoms in a multicenter study involving Italian ICUs. The proposal of the present study is to verify on a larger scale if these instruments can really ameliorate the empathic communication among staff members, without increase in workload, and to make less traumatic, for the family members, their experience during and after the ICU stay.

DETAILED DESCRIPTION:
Many recent studies described the comprehension, the satisfaction, and the psychological consequences due to the experience of an ICU admission of a loved one. Even if satisfaction about meetings and clinical information is about 90%, from 50 to 70% of family members reported an incomplete medical comprehension, and 70% showed symptoms of anxiety and depression. Many interventions may considerably improve their ICU experience, regarding both the comprehension and the emotions. For example, the family members of ICU patients that receive clear and reassuring information can deal better with the stress associated with their loved one illness, or may participate in the clinical decisional processes with awareness and lighter emotional distress.

Literature shows that relationship with families of ICU patients presents these problems:

1. comprehension of care essentials (diagnosis, prognosis about illness severity, interventions undertaken);
2. trust on ICU staff members;
3. management of their emotions (anxiety, fear, depression);
4. post-traumatic stress symptoms due to the concerns about life-threatening diseases of their loved one.

To ameliorate the relationship and the communication in the harsh ICU environment, and to meet the problems aforementioned, in 2012 some instruments for families were created (website, brochure, posters). They present in non-technical language the activities and the environment of ICU, with the aim to increase their comprehension and - at the same time - to make them feel not alone and powerless.

To evaluate the effectiveness of these information instruments, a before-and-after study was done in 2012 in 12 Italian ICUs. These instruments were demonstrated able to improve the correctness of communication about outcome and treatment (not about the illness and the organ dysfunctions, that is responsibility of local staff), and to decrease the post-traumatic symptoms. Anxiety and depression symptoms were showed non-significantly decreased. The physicians also reported an improvement in the quality of communication with families. (Intensive Care Med. 2017 Jan;43(1):69-79). The main study limitations were: low prevalence of internet browsing among families; few participating centers; lacking of complete diagnosis of PTSD, made after 6 months from traumatic event; lacking of characteristics of staff members who participated on the family meetings. The present larger, randomized and controlled trial was then designed, to replicate and verify the preliminary results, overcoming the limits and finding new strategies of communication.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* family member of ICU patient
* patient with mechanical ventilation length expected at admission > 48 hours;

Exclusion Criteria:

* refusal to participate;
* inability to understand Italian language;
* any previously diagnosed and not compensated psychiatric condition;
* absence of visiting relatives in the first 4 ICU days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Correctness of comprehension | 7 days
  Improvement in correctness of comprehension during the family meetings about medical information (main outcome: prognosis quo ad vitam), and about medical treatment and not diagnosis regarding organ dysfunction (comprehension assessment interview, CAI, minimum = 0, maximum = 16)

SECONDARY OUTCOMES:
Anxiety | 7 days
  Evaluation of anxiety on families after an ICU admission of a loved one (Hospital Anxiety and Depression Scale, HADS, for anxiety: minimum = 0, maximum = 21)
Depression | 7 days
  Evaluation of depression on families after an ICU admission of a loved one (Hospital Anxiety and Depression Scale, HADS, for depression: minimum = 0, maximum = 21)
Acute traumatic stress | 7 days
  Evaluation of traumatic experience (ICU admission of a loved one) influence on families in the early term of the first ICU week (short screening scale for symptoms of post-traumatic stress disorder, minimum = 0, maximum = 7)
Post-traumatic stress disorder | 6 months
  Evaluation of traumatic experience (ICU admission of a loved one) influence on families in the long term of 6 months after ICU discharge (PTSD check list for DSM V - civilian version, PCL-5, minimum = 0, maximum = 80)
Empathy | 2 months
  Evaluation of project effects on ICU staff involvement (Jefferson Scale for Physician Empathy, JSPE, minimum = 20, maximum = 140).
Burnout | 2 months
  Evaluation of project effects on work satisfaction in ICU staff members (Maslach burnout inventory, MBI, minimum = 0, maximum = 132).

CONTACTS AND LOCATIONS:
Locations (1):
- AO San Paolo - Polo Universitario, Milan, Italy

REFERENCES:
- [Result] Azoulay E, Chevret S, Leleu G, Pochard F, Barboteu M, Adrie C, Canoui P, Le Gall JR, Schlemmer B. Half the families of intensive care unit patients experience inadequate communication with physicians. Crit Care Med. 2000 Aug;28(8):3044-9. doi: 10.1097/00003246-200008000-00061. PMID 10966293
- [Result] Pochard F, Azoulay E, Chevret S, Lemaire F, Hubert P, Canoui P, Grassin M, Zittoun R, le Gall JR, Dhainaut JF, Schlemmer B; French FAMIREA Group. Symptoms of anxiety and depression in family members of intensive care unit patients: ethical hypothesis regarding decision-making capacity. Crit Care Med. 2001 Oct;29(10):1893-7. doi: 10.1097/00003246-200110000-00007. PMID 11588447
- [Result] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Result] Schwarzkopf D, Behrend S, Skupin H, Westermann I, Riedemann NC, Pfeifer R, Gunther A, Witte OW, Reinhart K, Hartog CS. Family satisfaction in the intensive care unit: a quantitative and qualitative analysis. Intensive Care Med. 2013 Jun;39(6):1071-9. doi: 10.1007/s00134-013-2862-7. Epub 2013 Feb 16. PMID 23417207
- [Result] Mistraletti G, Umbrello M, Mantovani ES, Moroni B, Formenti P, Spanu P, Anania S, Andrighi E, Di Carlo A, Martinetti F, Vecchi I, Palo A, Pinna C, Russo R, Francesconi S, Valdambrini F, Ferretti E, Radeschi G, Bosco E, Malacarne P, Iapichino G; http://www.intensiva.it Investigators. A family information brochure and dedicated website to improve the ICU experience for patients' relatives: an Italian multicenter before-and-after study. Intensive Care Med. 2017 Jan;43(1):69-79. doi: 10.1007/s00134-016-4592-0. Epub 2016 Nov 9. PMID 27830281
- [Derived] Mistraletti G, Mezzetti A, Anania S, Ionescu Maddalena A, Del Negro S, Giusti GD, Gili A, Iacobone E, Pulitano SM, Conti G, Bocci MG. Improving communication toward ICU families to facilitate understanding and reduce stress. Protocol for a multicenter randomized and controlled Italian study. Contemp Clin Trials. 2019 Nov;86:105847. doi: 10.1016/j.cct.2019.105847. Epub 2019 Sep 13. PMID 31525488